









# PARTICIPANT INFORMATION LEAFLET AND CONSENT FORM AIM 1

| TITLE OF RESEARCH PROJECT: | |
|---|---|
| TOTAL (Transmission of Tuberculosis Among Illicit drug use Linkages) | |
| DETAILS OF PRINCIPAL INVESTIGATOR (PI): | |
| Title, first name, surname: South Africa: Prof Robin Warren United States: Dr. Karen Jacobson | Ethics reference number: 11563 NCT04151602 |
| Full postal address: Faculty of Medicine and Health Sciences Stellenbosch University Francie van Zijl Drive, Tygerberg, 7505 | PI Contact number:<br>South African: +27 21 938 9251<br>Email US PI at kjacobso@bu.edu |

We would like to invite you to take part in a research project. Please take some time to read the information presented here, which will explain the details of this project. Please ask the study staff or doctor any questions about any part of this project that you do not fully understand. It is very important that you are completely satisfied that you clearly understand what this research entails and how you could be involved. Also, your participation is **entirely voluntary** and you are free to decline to participate. In other words, you may choose to take part, or you may choose not to take part. Nothing bad will come of it if you say no: it will not affect you negatively in any way whatsoever. Refusal to participate will involve no penalty or loss of benefits or reduction in the level of care to which you are otherwise entitled to. You are also free to withdraw from the study at any point, even if you do agree to take part initially.

This study has been approved by the **Health Research Ethics Committee at Stellenbosch University.** The study will be conducted according to the ethical guidelines and principles of the international Declaration of Helsinki, the South African Guidelines for Good Clinical Practice (2006), the Medical Research Council (MRC) Ethical Guidelines for Research (2002), and the Department of Health Ethics in Health Research: Principles, Processes and Studies (2015).

#### What is this research study all about?

PO Box 241, Cape Town, 8000

**South Africa** 

We are doing this research to understand if people who use drugs have been exposed to tuberculosis (TB), are at risk of developing TB disease, and how many have TB disease right now. We also want to know if having HIV, other substance use such as tobacco and alcohol, food insecurity, or depression affect those with TB disease. If you agree, you will be asked to sign this form, participate in a procedure called "sputum induction" where we will collect sputum samples from you for TB testing, provide a urine sample for drug testing, have your blood drawn, and have a portion of your visit recorded so we can count how many times you cough. You will also complete interviews that will ask about your substance use, health, social circle, and how you spend your time. We will also ask you to tell two of your friends about our study to see if they would want to also participate. If you decide to stay for the whole study you will attend 2 visits approximately one week from each other. You will find more information about what will happen in this study later in this form. If you are found to have TB we will ask you if you are interested in the second and third parts of the study. We will have a separate consent form for that and give you more details later if you are eligible.

#### Why do we invite you to participate?

If you are one of the first four people in our study, you were invited because you have previously reported to us that you use meth (tik) and/or Mandrax. If you are not one of the first four participants, you were invited to be in our study because you received a recruitment coupon from a peer who thought you may be eligible for our study.











#### What will your responsibilities be?

If you agree, you will be one of up to 800 people who will participate in this study. In this study, if you get diagnosed with TB or HIV you will not receive special treatment for your TB or HIV, but we will encourage, and transport, you to go to one of the clinics in Worcester for treatment. If you have any other health problems, you should seek medical care from a doctor or nurse.

If you choose to take part in the study, you will be asked to provide a fingerprint for identification, answer some questions about the use of drugs and other substances, your social network, and provide sputum, urine, and blood samples. We will also record a portion of your visit to count how many times you cough. You will be given two coupons to recruit other people who use drugs in your social circle.

You may be selected to take part in the second part of the study, for which you will be asked to give additional sputum samples and answer more questions about your daily activities and social contacts. You may also be selected to take part in the third part of the study, where you will be asked to spend part of a day at local clinic or hospital and have an x-ray taken, and a sample of your cough. You will have the option to participate, and if you want to, you will be given more details and will sign a separate consent form if you are selected for either of these parts of the study.

#### Screening visit

After you have read and signed the consent form, we will confirm that you are eligible to take part in the study. We will ask you to provide a fingerprint so we can confirm that you have not been in the study before, and we will use the results of your self-reported drug use and urine drug test. Depending on the results of the survey and the urine test, you may not be eligible to continue in the study. This part of the visit will take place in a location we have rented for the study and will take about 30 minutes.

#### **Enrolment visit**

The visit will take place at the same rented space in Worcester, ideally on the same day that you are screened. The study procedures should take up to 1.5 hours. At this visit, we will ask you to:

- Provide information on how we can contact and locate you
- Answer questions about yourself, medical conditions, and your tik/Mandrax, alcohol, tobacco, and other drug use
- Provide 15 ml (approximately 1. tbsp) blood to be tested for HIV, to check if your immune cells show higher risk for TB disease, and to see if you were ever exposed to COVID-19. You will not be given the results of this COVID-19 testing. This is not a test to determine if you are infected with the COVID-19 virus.
- You will be given your HIV test result and offered transport to the clinic for further care
- Provide 2 sputum samples to test for TB disease
- Answer questions about other people in your social circle who use drugs
- Have a portion of your visit audio recorded so we can count how many times you cough
- Receive up to two coupons that you can give to up to two people you know who use tik/Mandrax
  who would be interested to enroll in this study as well. You should only give the coupon(s) to peers
  who have never received coupons for our study before.

#### Follow-up visit

Everyone enrolled in this study will have a follow-up visit approximately one week, up to one month after their first visit. This visit should take about 30 minutes. We may collect additional information on your health from your medical records from one of the clinics in Worcester. At this visit, you will:

- Receive your sputum results from us and be referred and offered transport to the Worcester CDC or to your local clinic to start treatment if you have TB
- If your sputum samples are negative, be asked to provide up to 2 additional samples to retest for TB











- · Answer additional questions about drug use in your social circle
- Receive a voucher to the value of R50 for each participant (maximum two participants) who enrolled
  into the study with the recruitment coupon that you gave them, as long as they are a peer who
  never received a coupon before. If they came to us with a coupon before you will not receive R50
  for giving another coupon to that peer.

If we ask you to provide additional sputum for TB testing and it shows you may have TB, we will contact you to have you visit the study clinic for one additional visit where we will give you your TB results and link you to TB care.

If any sputum samples are positive for TB, the TB bacteria in your sputum may be sent to the United States for researchers to learn more about it.

We will also check with the clinic, the National Health Laboratory Services (NHLS) and/or the Western Cape Provincial Health Data Centre at the end of our study to see if you got sick with TB, HIV, or COVID-19 over the next 5 years, and if you were diagnosed with TB, HIV, or COVID-19, we will collect some information on your illness from those places. If you tell us you were ever in a SATVI study, we may contact SATVI to find out the name of the study you participated in and the treatment you received (if any).

#### Will you benefit from taking part in this research?

There is no direct benefit to you. If you take part in the study it will help us learn about how TB is spread in the community and if people who use drugs are affected by TB more than those who do not.

#### Are there any risks involved in your taking part in this research?

Participation in this study is voluntary. There are a few risks to you participating in the study.

- The urine test for drug use may cause some discomfort or distress. If you feel distressed by the results, we will ensure that you have access to services to help you cope.
- Blood draws may cause mild pain, bruising, bleeding, infection, and sometimes fainting. Our study nurses are trained properly to minimize such happenings.
- When we do the procedure to get sputum from you, you may experience discomfort. The main risks associated with the sputum procedure are nausea, vomiting, and feeling short of breath.
- There is a small chance of stigma. People may treat you differently if they know you are someone who uses drugs. The study team will do its best to keep your participation confidential, and each team member has to sign a confidentiality clause before starting on the project.
- You may feel uncomfortable by the personal nature of the guestions we will ask you.
- You may feel worried if you find out that you have TB and/or HIV, but we will link you to treatment at the local clinic to ensure that you start on treatment as soon as possible.
- We may store leftover samples that you provide us (blood and sputum) for studies that may not be
  planned yet for up to 10 years. While these samples will not have your name or any information
  about you, there is a small chance of breach of confidentiality.

If you feel stress from this study, you should tell our project staff. You can also take a break at any time. You have the right to stop participating in the study at any time, please tell our staff if you no longer want to continue.

#### If you do not agree to take part, what alternatives do you have?

Choosing to not take part in this study will not affect the medical care you receive anywhere at any time. If you have medical concerns you should seek out care at your preferred clinic.













#### Who will have access to your medical records?

Information from this study and from your medical records may be reviewed by the Stellenbosch University's (SU), SAMRC, and University of Cape Town (UCT) Research Ethics Committees and U.S. regulatory agencies such as the Office of Human Research Protection, the Institutional Review Board (IRB) of BMC and the NIH. Your contact information will be kept confidential and will be destroyed three years after the end of the study. Information from this study and your medical records may be used for research purposes and may be published. Your name will not be used in any publications.

To protect your privacy, information we collect from you will be stored with code numbers, rather than our name. A log that links your name to the code will be stored securely and will not be shared unless required by law. The fingerprint you provide will be scrambled and not stored as an image, so that no one will be able to access your unique fingerprint. If you enroll in TOTAL and then enroll in another study that uses the same fingerprint system that we use, the staff on that study may see that you are also enrolled in TOTAL but will not know any other information about you. Once TOTAL has been completed, we will remove you from the system so that you no longer show up as enrolled in TOTAL. Any studies who use this fingerprint system must sign an agreement that they will not share any information about who is enrolled in studies. The audio recording of your visit will be kept in a locked cabinet at Stellenbosch and will be destroyed up to one month after your coughs are counted. The laboratories processing your biological samples will never have access to your name. We will ask you at the end of this form if we can store your leftover samples (blood and sputum) at Stellenbosch University. We might use your research data/samples in future studies to help us understand more about tuberculosis and/or substance use. These future studies might be done by us or by other investigators but will never be for commercial purposes. Before we use your data/samples, we will remove any information that shows your identity. If you have concerns or questions about your stored specimens, you can contact the SU Health Research Ethics Committee at 021 938 9207.

This study is covered by a Certificate of Confidentiality (CoC) from the National Institutes of Health. All studies funded by the National Institutes of Health that involve identifiable information or biological samples are covered by a CoC. The CoC provides how we can share research samples or biological samples. Because we have a CoC, we cannot give out research information or biological samples that may identify you to anyone that is not involved in the research except as we describe below. Even if someone tries to get your information or biological samples in connection with a legal proceeding, we cannot give it to them. The CoC does not prevent you from sharing your own research information. The Certificate of Confidentiality applies to information and samples collected for this study which are sent to or kept in the United States of America.

Your information will be only be disclosed as required by law in the following two instances: 1) if you tell us that you are about to hurt yourself or someone else we will report this, or 2) if you are involved in the neglect or abuse of a child. We will then need to report that information to the authorities.

The information collected for this study, excluding your name and other contact information, will be stored at Stellenbosch University for at 15 years after the end of the study. Your specimens (blood and sputum) may be stored for up to 10 years.

## Even though it is unlikely, what will happen if you get injured somehow because you took part in this research study?

Stellenbosch University will provide comprehensive no-fault insurance and will pay for any medical cost that came about because participants took part in the research. The participant will not need to prove that the sponsor was at fault.

#### Will you be paid to take part in this study and are there any costs involved?

There is no cost for you to participate in this study. You will receive reimbursement in the form of grocery store vouchers to help cover your time, inconvenience, and expenses. You will receive a voucher to the value of R180 for the enrollment visit. There is the opportunity to receive an additional R100 (two R50 grocery vouchers) if you return for the follow up visit and have recruited two additional people into the study. These people should be someone who have not visited us before, and bring the coupon you gave them to the visit.

#### Is there anything else that you should know or do?

- ➤ You can phone the South African principal investigator, Prof Robin Warren at +27 21 938 9251, or email him at rw1@sun.ac.za. You can email the US principal investigator at kjacobso@bu.edu if you have any further queries or encounter any problems.
- ➤ You can phone the Health Research Ethics Committee at 021 938 9677/9819 if there still is something that your study doctor has not explained to you, or if you have a complaint.











> You will receive a copy of this information and consent form for you to keep safe.

| Declaration by part | ticipant |
|---|---|
| | agree to take part in a research study entitled f Tuberculosis Among Illicit drug use Linkages). |
| Please check <u>one</u> of the | options below (and initial): |
| (Participant initials) | I agree that my samples may be stored for up to 10 years after the study for use by the investigators on this study or other studies who are interested in learning more about tuberculosis and/ or substance use. |
| (Participant initials) | I do not agree to have my samples stored for use after the end of this study. |
| Please check one of the | options below (and initial): |
| (Participant initials) | I agree to be contacted after my time in the study by the investigators about matters related to this study or other potential studies I may be eligible for |
| (Participant initials) | I do not agree to be contacted after the study by investigators about matters related to this study or other potential studies I may be eligible for |
| I declare that: | |
| | s information and consent form, or it was read to me, and it is written in a ch I am fluent and with which I am comfortable. |
| <ul> <li>I have had a change answered.</li> </ul> | nance to ask questions and I am satisfied that all my questions have been |
| <ul> <li>I understand that<br/>take part.</li> </ul> | at taking part in this study is voluntary, and I have not been pressurised to |
| | o leave the study at any time and nothing bad will come of it – I will not be ejudiced in any way. |
| | to leave the study before it has finished, if the study doctor or researcher feels nterests, or if I do not follow the study plan that we have agreed on. |
| Signed at ( <i>place</i> ) | on ( <i>date</i> ) |
| Signature of participan | Signature of witness (if required) |

### Declaration by investigator/research staff member

I (name) ...... declare that:

- I explained the information in this document to ....., in a simple and clear manner
- I encouraged him/her to ask questions and took enough time to answer them.
- I am satisfied that he/she completely understands all aspects of the research, as discussed above.

BOSTON UNIVERSITY SCHOOLS OF MEDICINE, PUBLIC HEALTH, DENTAL MEDICINE AND THE BOSTON MEDICAL CENTER











• I did/did not use an interpreter. (If an interpreter is used then the interpreter must sign the declaration below.)

| Signature of investigator/research staff member | Signature of witness (if required) |
|---|---|
| Signed at (place) or | n ( <i>date</i> ) |